CLINICAL TRIAL: NCT04109755
Title: A Phase II Study to Evaluate Safety and Efficacy of Neo-adjuvant Pembrolizumab and Radiotherapy in Localised MSS Rectal Cancer
Brief Title: Neo-adjuvant Pembrolizumab and Radiotherapy in Localised MSS Rectal Cancer
Acronym: PEMREC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Thibaud Kossler, Medical Oncologist, University Hospital, Geneva
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEMREC
Record Dates: First submitted 2019-09-24; First posted 2019-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Rectum Cancer; Rectal Cancer
Keywords: Rectal cancer; Immunotherapy; Short course radiotherapy; 5x5Gy; Pembrolizumab; Localised rectal cancer
MeSH Terms: conditions — Rectal Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Short Course Radiation Therapy (5 x 5 Gy in 1 week, SCRT) with 4 injections of Pembrolizumab starting on the first day of radiotherapy and surgery
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 5x5 Gy radiotherapy in 1 week, 4 cycles of Pembrolizumab (200 mg every three week), surgery

SUMMARY:
This project investigates the clinical and biological impact of combining immunotherapy (pembrolizumab) with short course radiotherapy (5Gy, five times) in the neo-adjuvant treatment of localised microsatellite stable (MSS) rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male/female participants who are at least 18 years of age on the day of signing informed consent with histologically confirmed diagnosis of rectal adenocarcinoma will be enrolled in this study.
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the date of allocation.
* Patients with previously untreated localized T3-T4 N0 or T any or N1-2, M0 rectal adenocarcinoma.
* Tumour must be microsatellite stable (MSS).
* A multi-disciplinary tumour board should recommend neo-adjuvant short course radiotherapy and surgery.
* Have provided archival tumour tissue sample or newly obtained core or excisional biopsy of a tumour lesion not previously irradiated. Formalin-fixed paraffin embedded (FFPE) tissue blocks are preferred.
* Have adequate organ function as defined in the following table. Specimens must be collected within 10 days prior to the start of study treatment.

Exclusion Criteria:

* Has a microsatellite instable tumour (MSI-High).
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
* Has received for the same disease prior systemic anti-cancer therapy including investigational agents prior to starting pembrolizumab. Note: If participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
* Has received prior radiotherapy for the same disease. If treated with radiotherapy for another disease, participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
* Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment. Note: Participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has a known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded.
* Has known active CNS metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic therapy.
* Has a known history of Human Immunodeficiency Virus (HIV).
* Has a known history of Hepatitis B virus (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA > 1.5E1 is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-06-02 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Tumour regression grade | 12 weeks after start
  To assess the tumour regression grade (TRG) after short course radiotherapy when given together with pembrolizumab, using the Mandard regression grade score

SECONDARY OUTCOMES:
Tolerability and safety | 5 years
  To assess tolerability and safety of pembrolizumab given with short course radiotherapy before surgery, using the common terminology criteria for adverse events (CTCAE) Version 4.0
Overall Survival | 5 years
  To estimate overall survival (OS), defined as the time between the date of the study entry and the date of death due to any cause. Subjects who have not died at the time of last known follow-up will be censored.
Disease-free survival | 3 years
  To estimate disease-free survival (DFS), defined as the time between the date of the study entry and the date of recurrence, second primary cancer, or death without evidence of recurrence or second primary cancer.
Locoregional relapse-free survival | 5 years
  To estimate locoregional relapse-free survival (LRRFS), defined as the time between the date of the surgery and local or regional recurrence. LRRFS is evaluated in patients who had an R0 resection only
Distant metastasis-free survival | 5 years
  To estimate distant metastasis-free survival (DMFS), defined as the time between the date of the surgery and metastatic recurrence.
EORTC QLQ-C30 | 30 months
  European Organization for Research and Treatment of Cancer [EORTC] Quality of Life Questionnaire-C30
EORTC QLQ-CR29 | 30 months
  European Organization for Research and Treatment of Cancer [EORTC] Quality of Life Questionnaire-CR29

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Genève, Geneva, Switzerland

REFERENCES:
- [Derived] Corro C, Buchs NC, Tihy M, Durham-Faivre A, Bichard P, Frossard JL, Puppa G, McKee T, Roth A, Zilli T, Trembleau C, Di Marco M, Dutoit V, Dietrich PY, Ris F, Koessler T. Study protocol of a phase II study to evaluate safety and efficacy of neo-adjuvant pembrolizumab and radiotherapy in localized rectal cancer. BMC Cancer. 2022 Jul 15;22(1):772. doi: 10.1186/s12885-022-09820-w. PMID 35840912